CLINICAL TRIAL: NCT06791993
Title: Impact of Probiotics Combined with Antibiotic Prophylaxis on Gut Microbiome Balance in Patients Undergoing Elective Orthopedic Surgery, Double-Blinded Randomized Controlled Trial
Brief Title: Impact of Probiotics on Gut Microbiome During Antibiotic Prophylaxis in Elective Orthopedic Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Acibadem Maslak Hospital (Other)
Collaborators: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-KAEK-03
Record Dates: First submitted 2024-12-23; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Dysbiosis; Gut -microbiota; Microbiome Analysis; Probiotic; Antibiotic Prophylaxis
Keywords: Gut Microbiome; Intestinal Dysbiosis; Surgical Site Infection; Probiotics; Antibiotic Prophylaxis; Human Milk Oligosaccharides (HMO); Shotgun Metagenomic Sequencing; Short-Chain Fatty Acids (SCFAs)
MeSH Terms: conditions — Dysbiosis; Surgical Wound Infection | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This study uses a parallel group design where participants are randomly assigned to one of two independent arms. One group receives routine antibiotic prophylaxis with a placebo capsule, while the other group receives routine antibiotic prophylaxis combined with a dual-strain probiotic containing Human Milk Oligosaccharides (HMO). The interventions are administered concurrently over the perioperative period to evaluate their effects on gut microbiome balance and patient recovery. Randomization and blinding ensure unbiased comparisons between the groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In addition to participants, care providers, investigators, and outcomes assessors, the study's pharmacy personnel responsible for dispensing the intervention are also masked to the group assignments. Placebo and probiotic capsules are prepared to be identical in appearance and packaging, ensuring that no party involved in the trial can distinguish between the two interventions. Randomization and allocation are managed by an independent third party to maintain blinding integrity throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine Antibiotic Prophylaxis + Placebo (Placebo Comparator): This arm receives routine antibiotic prophylaxis with a single dose of intravenous Cefazolin and a placebo capsule to match the probiotic intervention.
  Interventions: Drug: Placebo Capsule
- Routine Antibiotic Prophylaxis + Probiotics (Experimental): This arm receives routine antibiotic prophylaxis with a single dose of intravenous Cefazolin and a dual-strain probiotic containing Human Milk Oligosaccharides (HMO).
  Interventions: Dietary Supplement: Probiotic with Human Milk Oligosaccharides (HMO)

INTERVENTIONS:
Drug: Placebo Capsule — Participants will receive an inert placebo capsule that matches the probiotic capsule in size, shape, and color. The placebo will be administered orally twice daily, starting 2 weeks before surgery and continuing for 2 weeks postoperatively.
  Arms: Routine Antibiotic Prophylaxis + Placebo
Dietary Supplement: Probiotic with Human Milk Oligosaccharides (HMO) — Participants will receive a dual-strain probiotic containing Human Milk Oligosaccharides (HMO) in capsule form. The probiotic will be administered orally twice daily, starting 2 weeks before surgery and continuing for 2 weeks postoperatively.
  Other Names: Dual-Strain Probiotic
  Arms: Routine Antibiotic Prophylaxis + Probiotics

SUMMARY:
This study aims to evaluate whether probiotics can help maintain a healthy gut microbiome in patients receiving prophylactic antibiotics during elective orthopedic surgery. Antibiotics, while effective in preventing infections, can disrupt the balance of gut bacteria, leading to dysbiosis. The study hypothesizes that the use of probiotics during the perioperative period can prevent or reduce this disruption, supporting gut health and overall well-being. The research seeks to answer whether combining probiotics with routine antibiotic prophylaxis can preserve gut microbiome balance and improve patient outcomes.

DETAILED DESCRIPTION:
This double-blinded, randomized controlled trial aims to evaluate the effect of probiotics on maintaining gut microbiome balance in patients undergoing elective orthopedic surgery who receive routine prophylactic antibiotics. Antibiotics, while essential for reducing the risk of surgical site infections, are known to disrupt gut microbiota, leading to dysbiosis, an imbalance in microbial composition. Dysbiosis can compromise gut health, reduce microbial diversity, and impair metabolic functions essential for recovery.

The study explores whether a dual-strain probiotic with Human Milk Oligosaccharides (HMO) can prevent or minimize dysbiosis during the perioperative period. By comparing patients receiving routine antibiotics alone with those receiving antibiotics plus probiotics, this trial seeks to identify if probiotics can preserve gut microbial diversity and function.

To assess the impact, fecal samples collected at specific time points will undergo detailed microbiome analysis, including metrics such as microbial richness, diversity, and such. Secondary measures will evaluate the broader effects on patient well-being during the recovery period.

This study is designed to provide evidence for the potential role of probiotics as an adjunct therapy to maintain gut health during antibiotic use, offering a novel approach to improving post-surgical recovery and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years
* Scheduled for elective low-risk orthopedic surgery (carpal tunnel release, A1 pulley release, knee arthroscopic surgery).

Exclusion Criteria:

* History of infection or antibiotic use within the last 12 weeks.
* Use of routine probiotics, vitamins, or herbal supplements in the last 4 weeks.
* Known allergy to beta-lactam or cephalosporin antibiotics.
* History of autoimmune disease, uncontrolled systemic disease, or chronic inflammatory conditions (e.g., systemic lupus erythematosus, rheumatoid arthritis).
* History of chronic intestinal diseases such as small intestine bacterial overgrowth (SIBO), irritable bowel syndrome (IBS), inflammatory bowel disease (IBD), or celiac disease.
* Increased risk of infection due to medical comorbidities or use of immunosuppressive drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Maintenance of Gut Microbiome Balance | 2 weeks preoperatively (T0) to 1 month postoperatively (T4).
  Evaluate whether probiotic administration preserves gut microbiome balance during the perioperative period by assessing changes in microbial richness, diversity, and evenness. Shotgun metagenomic sequencing analysis will be used to measure microbial composition and diversity.

SECONDARY OUTCOMES:
Firmicutes/Bacteroidetes Ratio | 2 weeks preoperatively (T0) to 1 month postoperatively (T4).
  Determine changes in the Firmicutes/Bacteroidetes ratio, a key marker of dysbiosis, between intervention groups. Using shotgun metagenomic sequencing.
Short-Chain Fatty Acid (SCFA) Production | 2 weeks preoperatively (T0) to 1 month postoperatively (T4).
  Assess changes in SCFA production (e.g., acetate, butyrate) as indicators of gut health and microbiome function. Using SCFA quantification through microbiome metabolite analysis.
Dysbiosis Index | 2 weeks preoperatively (T0) to 1 month postoperatively (T4).
  Dysbiosis Index is the ratio of the total number of Proteobacteria strains divided by total overall bacteria strain
Microbiome health index ( MHI) OR Microbiome health index for post-antiobiotic (MHI- A) | 2 weeks preoperatively (T0) to 1 month postoperatively (T4).
  Microbiome Health Index (MHI-A) calculated via microbiome analysis. MHI-A is a biomarker and a quantitative measure method of post-antibiotic dysbiosis and subsequent restoration. Higher MHI-A means higher healthy microbiome with low antibiotic resistance gene. Lower MHI- A mean dysbiosis, high antiobiotic resistance gene
WHO-5 Well-being Index | 1 week preoperatively (T1) and 2 weeks postoperatively (T3).
  The WHO-5 Well-Being Index (The World Health Organization-Five Well-Being Index) is a self-report instrument measuring mental well-being. It consists of five statements relating to the past two weeks. Each statement is rated on a 6-point scale (0,1,2,3,4,5), with higher scores indicating better mental well-being.
  The raw score is calculated by totalling the scores on each of the five questions. Theraw score ranges from zero to 25, zero representing worst possible mental well-beingand 25 representing best possible mental well-being. To get a percentage score ranging from zero to 100, the raw score is multiplied by four.
  A percentage score of zero represents worst possible mental well-being; a score of 100 represents best possible mental well-being
EuroQol 5-Dimension (EQ-5D) score. | 1 week preoperatively (T1) and 2 weeks postoperatively (T3).
  EuroQol 5-Dimension (EQ-5D) score (EQ-5D) descriptive system comprises the same five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION), beach dimension having five response levels:no problems, slight problems, moderateproblems, severe problems, unable to/extreme problems. The respondent is asked to indicate his/her health state by checking the box next to the most appropriate response level for each of the five dimensions. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the five dimensions can be combined in a 5-digit code that describes the respondent's health state; for instance, 21111 means slight problems in the mobility dimension and no problems in any of the other dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Javad Parvizi, Prof. Dr., Study Chair — International Joint Center Acibadem, Parvizi Surgical Innovation; Emanuele Chisari, Dr., Ph.D., Study Director — Parvizi Surgical Innovation, University of Groningen
Locations (6):
- Parvizi Surgical Innovation, Philadelphia, Pennsylvania, United States
- Thonburi Trang Hastanesi, Thailand, Thailand
- Turkey (Türkiye) (4):
  - Istanbul University Cerrahpasa, Istanbul
  - Acıbadem International Joint Center, Istanbul
  - Acibadem LABMED Laboratories, Istanbul
  - Acıbadem Mehmet Ali Aydınlar University, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Data access will be granted to researchers who provide a methodologically sound proposal. Proposals should be directed to goksel.dikmen@acibadem.com To gain access, data requestors will need to sign a data access agreement.
URL: https://www.drive.google.com/drive/folders/1C-CfBwEXCHEXl86ePRO4o4opAShsa9Op?usp=drive_link

REFERENCES:
- [Background] Anthony WE, Wang B, Sukhum KV, D'Souza AW, Hink T, Cass C, Seiler S, Reske KA, Coon C, Dubberke ER, Burnham CD, Dantas G, Kwon JH. Acute and persistent effects of commonly used antibiotics on the gut microbiome and resistome in healthy adults. Cell Rep. 2022 Apr 12;39(2):110649. doi: 10.1016/j.celrep.2022.110649. PMID 35417701
- [Background] Rios JL, Bomhof MR, Reimer RA, Hart DA, Collins KH, Herzog W. Protective effect of prebiotic and exercise intervention on knee health in a rat model of diet-induced obesity. Sci Rep. 2019 Mar 7;9(1):3893. doi: 10.1038/s41598-019-40601-x. PMID 30846801
- [Background] Akagawa Y, Kimata T, Akagawa S, Yamaguchi T, Kato S, Yamanouchi S, Hashiyada M, Akane A, Kino M, Tsuji S, Kaneko K. Impact of Long-Term Low Dose Antibiotic Prophylaxis on Gut Microbiota in Children. J Urol. 2020 Dec;204(6):1320-1325. doi: 10.1097/JU.0000000000001227. Epub 2020 Jul 2. PMID 32614253
- [Background] Huang Z, Chen J, Li B, Zeng B, Chou CH, Zheng X, Xie J, Li H, Hao Y, Chen G, Pei F, Shen B, Kraus VB, Wei H, Zhou X, Cheng L. Faecal microbiota transplantation from metabolically compromised human donors accelerates osteoarthritis in mice. Ann Rheum Dis. 2020 May;79(5):646-656. doi: 10.1136/annrheumdis-2019-216471. Epub 2020 Mar 23. PMID 32205337
- [Background] Coulson S, Butt H, Vecchio P, Gramotnev H, Vitetta L. Green-lipped mussel extract (Perna canaliculus) and glucosamine sulphate in patients with knee osteoarthritis: therapeutic efficacy and effects on gastrointestinal microbiota profiles. Inflammopharmacology. 2013 Feb;21(1):79-90. doi: 10.1007/s10787-012-0146-4. Epub 2012 Jul 22. PMID 22821424
- [Background] Kullar R, Chisari E, Snyder J, Cooper C, Parvizi J, Sniffen J. Next-Generation Sequencing Supports Targeted Antibiotic Treatment for Culture Negative Orthopedic Infections. Clin Infect Dis. 2023 Jan 13;76(2):359-364. doi: 10.1093/cid/ciac733. PMID 36074890
- [Background] Ramires LC, Santos GS, Ramires RP, da Fonseca LF, Jeyaraman M, Muthu S, Lana AV, Azzini G, Smith CS, Lana JF. The Association between Gut Microbiota and Osteoarthritis: Does the Disease Begin in the Gut? Int J Mol Sci. 2022 Jan 27;23(3):1494. doi: 10.3390/ijms23031494. PMID 35163417
- [Background] Chisari E, Wouthuyzen-Bakker M, Friedrich AW, Parvizi J. The relation between the gut microbiome and osteoarthritis: A systematic review of literature. PLoS One. 2021 Dec 16;16(12):e0261353. doi: 10.1371/journal.pone.0261353. eCollection 2021. PMID 34914764
- [Background] Favazzo LJ, Hendesi H, Villani DA, Soniwala S, Dar QA, Schott EM, Gill SR, Zuscik MJ. The gut microbiome-joint connection: implications in osteoarthritis. Curr Opin Rheumatol. 2020 Jan;32(1):92-101. doi: 10.1097/BOR.0000000000000681. PMID 31724973
- [Background] Boer CG, Radjabzadeh D, Medina-Gomez C, Garmaeva S, Schiphof D, Arp P, Koet T, Kurilshikov A, Fu J, Ikram MA, Bierma-Zeinstra S, Uitterlinden AG, Kraaij R, Zhernakova A, van Meurs JBJ. Intestinal microbiome composition and its relation to joint pain and inflammation. Nat Commun. 2019 Oct 25;10(1):4881. doi: 10.1038/s41467-019-12873-4. PMID 31653850
- See also: Related Info — https://drive.google.com/drive/folders/1C-CfBwEXCHEXl86ePRO4o4opAShsa9Op
- Available data/document: Individual Participant Data Set — https://drive.google.com/drive/folders/1C-CfBwEXCHEXl86ePRO4o4opAShsa9Op — https://drive.google.com/drive/folders/1C-CfBwEXCHEXl86ePRO4o4opAShsa9Op